CLINICAL TRIAL: NCT00313846
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Determine the Efficacy and Safety of the Buprenorphine Transdermal Delivery System in Subjects With Moderate to Severe Osteoarthritic Pain of Hip or Knee
Brief Title: Safety and Efficacy of Buprenorphine Transdermal System in Subjects With Moderate to Severe Osteoarthritis of Hip or Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUP3012
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Results first posted 2010-09-28 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Osteoarthritis
Keywords: Chronic pain; opioid; transdermal; osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Chronic Pain | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- BTDS (Experimental): Buprenorphine transdermal patch 5, 10 or 20 micrograms/hour (mcg/h)
  Interventions: Drug: Buprenorphine transdermal patch
- Placebo (Placebo Comparator): Placebo to match BTDS 5, 10 or 20 mcg/h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 5, 10 or 20 mcg/h applied for 7-day wear.
  Other Names: Butrans™
  Arms: BTDS
Drug: Placebo — Placebo to match BTDS 5, 10, or 20 mcg/h applied for 7-day wear.
  Arms: Placebo

SUMMARY:
The objective of this study is to demonstrate the effectiveness and tolerability of the buprenorphine transdermal system (BTDS) (5, 10 and 20) in comparison to placebo transdermal system in subjects with moderate to severe osteoarthritis pain of the hip and knee currently treated with oral opioids. The double-blind treatment intervention duration is 4 weeks during which time supplemental analgesic medication (acetaminophen) will be provided to all subjects in addition to study drug.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over 25 years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of chronic osteoarthritis of the hip or knee for 1 year or longer.
* an average pain due to osteoarthritis of moderate, moderately-severe, or severe for the 14 days prior to enrollment.

Exclusion Criteria:

* ingest opioid analgesics on a daily basis.
* ingest >2500 milligrams (mg) acetaminophen on a daily basis.
* require <20 mg or >80 mg of morphine (or opioid equivalents) per day for control of their osteoarthritis pain.

Other protocol-specific exclusion/inclusion criteria may apply.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2003-04; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - Vista Medical Research, Mesa, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Radiant Research, Phoenix, Arizona
  - ACRC/Arizona Clinical Research, Tucson, Arizona
  - Advance Pain Medicine, Bakersfield, California
  - Eastgate Medical Center, Cypress, California
  - University Osteoporosis Ctr, Loma Linda, California
  - San Diego Arthritis & Osteoporosis Medical Clinic, San Diego, California
  - Scripps Clinic Rancho Bernard, San Diego, California
  - CNS Clinical Trials, Inc, San Francisco, California
  - Mountain View Clinical Research, Denver, Colorado
  - Integrative Treatment Centers/Rocky Mtn Clin Res, Westminster, Colorado
  - Rocky Mountain Center for Clinical Research, Wheat Ridge, Colorado
  - Stamford Therapeutic Consortium, Bridgeport, Connecticut
  - Medical Specialists of the Palm Beaches, Atlantis, Florida
  - University Clinical Research Deland, DeLand, Florida
  - Drug Study Institute, Jupiter, Florida
  - Coastal Medical Research, Orange City, Florida
  - Coastal Medical Research, Port Orange, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Gold Coast Research, Weston, Florida
  - Non-Surgical Orthopedic & Spine Center, Marietta, Georgia
  - Columbus Internal Medical Associates, Columbus, Indiana
  - MediSphere Medical Research Ctr., Evansville, Indiana
  - Primary Care Research, Murray, Kentucky
  - Professional Clinical Research, Cadillac, Michigan
  - Sound Medical At West Front Primary Care, Traverse City, Michigan
  - Beth Israel Med Ctr Dept of Pain Medicine & Palliative Care, New York, New York
  - All-Trials Clinical Research, LLC, Winston-Salem, North Carolina
  - Keystone Clinical, Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Clinical Research Center of Reading, LLP, West Reading, Pennsylvania
  - Low Country Rheumatology, Charleston, South Carolina
  - Brown Clinic, Watertown, South Dakota
  - Private Practice, Dallas, Texas
  - Team Research of Central Texas, Harker Heights, Texas
  - Radiant Research San Antonio Northeast, San Antonio, Texas
  - ACCU Clinical Research Trials, Inc, Seguin, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Advance Pain Management & Rehab, Virgina Beach, Virginia
  - Evergreen Clinical Research Associates, Edmonds, Washington
  - Internal Medicine Northwest, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25-Apr-2003 (first patient first visit) to 01-Jun-2004 (last patient last visit).
  This study was conducted at 41 medical/research sites in the United States.
Pre-assignment Details: 529 subjects began the run-in period with buprenorphine transdermal system (BTDS) 5 and their dose was titrated to BTDS 10 or 20 to achieve effective pain control. Subjects meeting criteria for adequate analgesia within 21 days were randomized into the double-blind phase (the number of subjects [N] = 328 completed run-in period).
Groups:
- Double-blind Placebo: Reference treatment in the double-blind phase. Placebo transdermal patches matched the BTDS patches applied for 7-day wear.
- Double-blind BTDS: Test treatment in the double-blind phase. Buprenorphine transdermal patches 5, 10, or 20 applied for 7-day wear.
Period: Overall Study
Arm/Group | Double-blind Placebo | Double-blind BTDS
Started | 162 | 164 (327 subjects were randomized: 1 subject was lost to follow-up (N = 326).)
Completed | 157 | 153
Not Completed | 5 | 11
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 1 | 8
Not completed — Administrative | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind Placebo | Double-blind BTDS | Total
Number analyzed (Participants) | 162 | 164 | 326
Age Continuous [Mean (Standard Deviation); unit: years] | 61.2 (9.64) | 60.4 (9.28) | 60.8 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 113 | 219
  Male | 56 | 51 | 107

OUTCOME MEASURES:

1. Primary Outcome: The Time (Days) From First Administration of Double-blind Treatment to the Development of Inadequate Analgesia at the Primary Osteoarthritis Pain Site.
Description: Inadequate analgesia:
  * "average pain over the last 24 hours" score for pain at primary osteoarthritis (OA) site ≥ 5 on any 2 days of any 7-day dosing period, on a scale from 0 - 10 (0 = no pain to 10 = pain as bad as you can imagine)or;
  * >1000 mg/day acetaminophen for pain at primary OA site for ≥ 2 days in any 7-day dosing period, or;
  * ingested nonstudy opioid analgesic medication for pain at primary OA site. Score: lowest score = shortest time to inadequate analgesia; highest score = longest time to inadequate analgesia.
Time Frame: Double-blind phase ( 28 days): reaching "inadequate analgesia" on any 2 days of the 7-day dosing periods
Population: The Full Analysis Population (N = 326) consisted of subjects who were randomized and received at least 1 dose of double-blind study drug and had at least 1 primary efficacy observation during the double-blind phase.
Measure: Mean (Standard Error); unit: days
Arm/Group | Double-blind Placebo | Double-blind BTDS
Number analyzed (Participants) | 162 | 164
days | 12.3 (0.77) | 17.2 (0.89)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind BTDS; Test type: Superiority or Other; p = .0026, Kaplan-Meier estimate mean

2. Secondary Outcome: Daily Maximum "Pain Right Now" Score for the Primary Osteoarthritis (OA) Pain Site
Description: The daily maximum 'pain right now' score for the primary OA pain site was calculated over the last 7-day dosing period in the double-blind phase or the last 7-day dosing period prior to emergence of inadequate analgesia or discontinuation from the double-blind phase. Collected prior to ingestion of acetaminophen. "Pain right now" scale score for primary OA site on a scale from 0-10 (where 0= no pain and 10= worst pain you can imagine).
Time Frame: 7 days of the last dosing period of the double-blind phase, or the last 7-day dosing period prior to emergence of inadequate analgesia or discontinuation from the double-blind phase.
Population: Full Analysis Population (N = 326) consisted of subjects who were randomized and received at least 1 dose of double-blind study drug and had at least 1 primary efficacy observation during the double-blind phase.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind Placebo | Double-blind BTDS
Number analyzed (Participants) | 162 | 164
units on a scale | 3.8 (0.15) | 3.2 (0.14)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) that occurred after the signing of the informed consent up to end of study and 7 days after, or discontinuation, or Serious AEs occurring up to 30 days following the last study visit were followed until the AE resolved or stabilized.
Description: Adverse events (AEs) were recorded through spontaneous reports and subject interview.
Groups:
- Double-blind Placebo Patch 5, 10, or 20: Reference treatment in the double-blind phase
- Double-blind BTDS 5, 10, or 20: Test treatments in the double-blind phase
- Open-label Run-in Period BTDS 5, 10, or 20: Open-label Run-in Period (less than or equal to 21 days): All subjects began treatment on BTDS 5 and titrated to a maximum of BTDS 20 to achieve effective pain control. Subjects were treated for a minimum of 3 days with any given dose of BTDS before up-titration to the next strength patch was considered. One down-titration was permitted. Subjects meeting protocol-defined criteria for adequate analgesia within 21 days were eligible for entry into the double-blind phase.
Arm/Group | Double-blind Placebo Patch 5, 10, or 20 | Double-blind BTDS 5, 10, or 20 | Open-label Run-in Period BTDS 5, 10, or 20
Serious Adverse Events (participants affected / at risk) | 0/162 | 1/164 | 6/529
Other Adverse Events (participants affected / at risk) | 15/162 | 28/164 | 229/529
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Placebo Patch 5, 10, or 20 (N=162) | Double-blind BTDS 5, 10, or 20 (N=164) | Open-label Run-in Period BTDS 5, 10, or 20 (N=529)
Intermittent complete heart block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Left foot cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Acute upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Elevated blood pressure (Investigations) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Transient ischemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessment
Numbness left side of face (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessment
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Tremulousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
Worsening of hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessment
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo Patch 5, 10, or 20 (N=162) | Double-blind BTDS 5, 10, or 20 (N=164) | Open-label Run-in Period BTDS 5, 10, or 20 (N=529)
Nausea (Gastrointestinal disorders) | 3 | 12 | 113 — Systematic and nonsystematic assessment
Constipation (Gastrointestinal disorders) | 6 | 10 | 41 — Systematic and nonsystematic assessment
Vomiting not otherwise specified (NOS) (Gastrointestinal disorders) | 0 | 1 | 36 — Systematic and nonsystematic assessment
Application site erythema (General disorders) | 5 | 9 | 6 — Systematic and nonsystematic assessment
Application site pruritus (General disorders) | 4 | 8 | 28 — Systematic and nonsystematic assessment
Headache (Nervous system disorders) | 15 | 7 | 65 — Systematic and nonsystematic assessment
Dizziness (Nervous system disorders) | 4 | 5 | 55 — Systematic and nonsystematic assessment
Somnolence (Nervous system disorders) | 0 | 2 | 41 — Systematic and nonsystematic assessment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days